CLINICAL TRIAL: NCT02556177
Title: Advanced MRI Applications for Mild Traumatic Brain Injury-Phase 2
Acronym: mTBI-phase2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GE Healthcare (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 114-2015-GES-0017
Record Dates: First submitted 2015-08-07; First posted 2015-09-22 (Estimated); Results first posted 2019-09-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Concussion; Traumatic Brain Injury
Keywords: TBI; MR; mTBI; NFL; MRI
MeSH Terms: conditions — Brain Concussion; Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- mTBI patient group (Segment 1) (Active Comparator): 1.5T or 3.0T MRI brain scanning with research sequences at 3 to 4 intervals in the acute period, with psychological cognitive evaluations at each MR visit
  Patients in the acute period following recent diagnosis of mild traumatic brain injury (mTBI)
  Interventions: Procedure: MRI
- non-TBI patients (Segment 2) (Active Comparator): Control subjects with no recent mild traumatic brain injury. 1.5T or 3.0T MRI brain scanning with research sequences at 3 to 4 intervals in the acute period, with psychological cognitive evaluations at each MR visit
  Interventions: Procedure: MRI

INTERVENTIONS:
Procedure: MRI — MRI scanning

SUMMARY:
This is an open-label, non-randomized, prospective, multi-site, parallel group (segment), hypothesis-generating study designed to collect data that will aid in future scientific and engineering exploration of correlations between clinical neuropsychological assessments and GE Research Pack II advanced MR imaging in mTBI patients. The results are primarily intended for scientific inquiry and engineering development purposes, and may be used in future regulatory submissions.

DETAILED DESCRIPTION:
This data-driven study is being conducted for hypothesis generation in population of mild traumatic brain injury (mTBI) patients using advanced applications for magnetic resonance imaging (MRI) developed by the Sponsor, GE Healthcare (GEHC), and corresponding clinical neuropsychological assessments. This data is intended for future use in development of specialized MR acquisition, reconstruction, and processing software intended to identify mTBI biomarkers.

ELIGIBILITY:
Inclusion Criteria:

Subjects included as mTBI patients (Segment 1) will:

1. Be aged ≥15 and ≤50 years old at the time of enrollment;
2. Be diagnosed with mTBI according to the standard diagnostic procedures at the investigational site in a timeframe that meets enrollment criteria for enrollment within 72 hours (Visit 1) or 7±2 days (Visit 3) from injury.
3. Be capable of sufficiently clear communication and language fluency to allow the subject to provide written informed consent, or assent with parental or guardian consent for minors, and to complete study assessments (as per Section 6.3 - Protection of Vulnerable Subjects) for participation in all parts of the study.

Subjects included as non-mTBI controls (Segment 2) will:

1. Be aged ≥15 and ≤50 years old at the time of enrollment;
2. Are of similar characteristics as the mTBI population in terms of gender, age, handedness, educational level, and scanner criteria (as per Section 6.1.1 Enrollment of non-mTBI controls)
3. Be capable of sufficiently clear communication and language fluency to allow the subject to provide written informed consent, or assent with parental or guardian consent for minors, and to complete study assessments (as per Section 6.3 - Protection of Vulnerable Subjects), for participation in all parts of the study.

Exclusion Criteria:

Subjects will be excluded that have: mTBI

1. Loss of consciousness (LOC) ≥5 minutes;
2. Posttraumatic amnesia lasting ≥24 hr following mTBI;
3. Current or prior (within past 10 years) moderate to severe TBI
4. Diagnosis of mTBI within the past 6 months;
5. Epilepsy with recurring seizures in past 10 years;
6. Drug abuse (except marijuana) in past 10 years based on DAST-10 screening;
7. Alcohol abuse based on AUDIT-C screening;
8. Current primary Axis I or II psychiatric disorders, except for disorders classified as minor and not expected to impact study conduct or integrity (as detailed in Appendix C - Screening Axis I/II Disorders):
9. History of brain mass, neurosurgery, stroke, white matter disease, and/or dementia;
10. Known cognitive dysfunction or structural brain disease/malformation;
11. Structural brain injury on prior neuroimaging findings;
12. Been prescribed antipsychotic/antiepileptic medications;
13. Unable (such as due to urgent medical care needs) or unwilling to complete study procedures accurately or have any conflict of interest that could affect study results, in the opinion of the investigator;
14. Contraindications to MRI scanning, including:

    * Current or suspected pregnancy, per site practice;
    * Other conditions that may constitute a hazard to the subject during study participation, per investigator;
    * Inability to comply with any part of the site's MR safety policy.

Subjects will be excluded that have:- non-TBI (controls)

1. Diagnosis of mTBI within the past 6 months;
2. Prior (within past 10 years) moderate to severe TBI (GCS <13);
3. Epilepsy with recurring seizures in past 10 years;
4. Drug abuse (except marijuana) in past 10 years based on DAST-10 screening;
5. Alcohol abuse based on AUDIT-C screening;
6. Current primary Axis I or II psychiatric disorders, except for disorders classified as minor and not expected to impact study conduct or integrity (as detailed in Appendix C - Screening Axis I/II Disorders):
7. History of brain mass, neurosurgery, stroke, white matter disease, and/or dementia;
8. Known cognitive dysfunction or structural brain disease/malformation;
9. Structural brain injury on prior neuroimaging findings;
10. Been prescribed antipsychotic/antiepileptic medications;
11. Unable (such as due to urgent medical care needs) or unwilling to complete study procedures accurately or have any conflict of interest that could affect study results, in the opinion of the investigator;

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 477 (Actual)
Dates: Start 2015-11; Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victor Miranda, MD, Study Director — GE Healthcare
Locations (7):
- United States (7):
  - University of California-San Diego, San Diego, California
  - University of California San Francisco, San Francisco, California
  - Universtiy of Miami Health System, Miami, Florida
  - Hospital for Special Surgery, New York, New York
  - University of Pittsburgh Medical College, Pittsburgh, Pennsylvania
  - Houston Methodist Neurological Institute, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Tanwar M, Miller E, Tsiouris AJ, Nguyen J, Agarwal V, Marinelli L, Erdemir GA, Shetty T. White Matter Hyperintensities on High-Resolution 3-T MRI: Frequency in Mild Traumatic Brain Injury and Associations With Clinical Markers-A Prospective Controlled Multicenter Study. AJR Am J Roentgenol. 2025 May;224(5):e2432274. doi: 10.2214/AJR.24.32274. Epub 2025 Feb 19. PMID 39969142

RESULTS

PARTICIPANT FLOW:
Groups:
- mTBI Patient Group (Segment 1): 1.5T or 3.0T MRI brain scanning with research sequences at 3 to 4 intervals in the acute period, with psychological cognitive evaluations at each MR visit
  Patients in the acute period following recent diagnosis of mild traumatic brain injury (mTBI)
  MRI: MRI scanning
Period: Overall Study
Arm/Group | mTBI Patient Group (Segment 1) | Non-TBI Patients (Segment 2)
Started | 325 | 152
Completed | 42 | 91
Not Completed | 283 | 61
Not completed — Subjects did not complete all 4 visits | 283 | 61

BASELINE CHARACTERISTICS:
Population: Segment 1 consisted of adolescent and adult mTBI patients who recently sustained head injury. Segment 2 consisted of subjects who were enrolled as a control population.
Groups:
- Total: Total of all reporting groups
Arm/Group | mTBI Patient Group (Segment 1) | Non-TBI Patients (Segment 2) | Total
Number analyzed (Participants) | 325 | 152 | 477
Age, Categorical [Count of Participants; unit: Participants] — Population: 8 subjects in Segment 1 did not collect age, as a result the overall subjects to be counted for age is 317.
  13 subjects in Segment 2 did not collect age, as a result the overall subjects to be counted for age is 139.
  Participants
    number analyzed (Participants) | 317 | 139 | 456
    <=18 years | 168 | 76 | 244
    Between 18 and 65 years | 149 | 63 | 212
    >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 8 subjects in Segment 1 did not collect gender, as a result the overall subjects to be counted for gender is 317.
  13 subjects in Segment 2 did not collect gender, as a result the overall subjects to be counted for gender is 139.
  Participants
    number analyzed (Participants) | 317 | 139 | 456
    Female | 141 | 76 | 217
    Male | 176 | 63 | 239
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 325 | 152 | 477

OUTCOME MEASURES:

1. Primary Outcome: MRI Image Data Sets
Description: MRI image data sets collected from subjects who completed the study.
Time Frame: Per patient scanning over 3 months
Measure: Number; unit: Images collected
Arm/Group | mTBI Patient Group (Segment 1) | Non-TBI Patients (Segment 2)
Number analyzed (Participants) | 325 | 152
Images collected
  Study Visit 1 images collected | 79 | 150
  Study Visit 2 images collected | 290 | 111
  Study Visit 3 images collected | 240 | 105
  Study Visit 4 images collected | 218 | 118
  Total number of images collected | 827 | 484

2. Primary Outcome: Neuropsychological Assessments
Description: Neuropsychological assessments collected from subjects who completed the study.
Time Frame: Per patient scanning over 3 months
Measure: Number; unit: Neuropsychological assessments
Arm/Group | mTBI Patient Group (Segment 1) | Non-TBI Patients (Segment 2)
Number analyzed (Participants) | 325 | 152
Neuropsychological assessments
  Visit 1 Neuropsychological assessments | 84 | 152
  Visit 2 Neuropsychological assessments | 303 | 114
  Visit 3 Neuropsychological assessments | 244 | 107
  Visit 4Neuropsychological assessments | 222 | 119
  Total number of Neuropsychological assessments | 853 | 492

ADVERSE EVENTS:
Time Frame: Each visit lasted approximately 90 minutes.
Description: Subjects were followed for adverse events and device effects from the time they arrived for each study visit (immediately after providing informed consent for the first visit, and upon arriving to the study area for each subsequent visit,) until the subject left the study area after each visit.
Arm/Group | mTBI Patient Group (Segment 1) | Non-TBI Patients (Segment 2)
All-Cause Mortality (participants affected / at risk) | 0/325 | 0/152
Serious Adverse Events (participants affected / at risk) | 0/325 | 0/152
Other Adverse Events (participants affected / at risk) | 22/325 | 1/152
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | mTBI Patient Group (Segment 1) (N=325) | Non-TBI Patients (Segment 2) (N=152)
Peripheral Nerve Stimulation (Nervous system disorders) | 5 (5) | 0 (0)
Claustrophobia (Nervous system disorders) | 7 (7) | 1 (1)
Headache (General disorders) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 3 (3) | 0 (0) — Pain and discomfort
Concussion (Nervous system disorders) | 3 (3) | 0 (0)
ACL tear (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Participant tore her ACL playing football between visits 3 and 4. Had surgery to repair.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-14): https://cdn.clinicaltrials.gov/large-docs/77/NCT02556177/Prot_SAP_000.pdf